CLINICAL TRIAL: NCT03111290
Title: Modulating Oscillations and Working Memory in Patients With Subdural Electrodes
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-2710; 1R21NS094988 (NIH); 1R01MH124387 (NIH)
Record Dates: First submitted 2017-02-22; First posted 2017-04-12 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Working Memory; Epilepsy
Keywords: Facial recognition
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (Sham Comparator): Device: Direct Cortical Stimulation Sham. Trials in which stimulation is not applied. These trials are initiated using a generic trigger generator.
  Interventions: Device: Direct Cortical Stimulation Sham
- Stimulation (Active Comparator): Device: Direct Cortical Stimulation. 150 stimulations with stimulations lasting 5 seconds at different target electrodes at two target frequencies (e.g. 5 Hz and 10 Hz) 2 milliampere in amplitude (Pulse shape - Biphasic square pulse 200 microsecond in duration per phase). Stimulation will be applied concurrently with the task and stimulation trials will be randomly interleaved with sham trials.
  Interventions: Device: Direct Cortical Stimulation

INTERVENTIONS:
Device: Direct Cortical Stimulation — A train of periodic electrical pulses is delivered between two local electrodes implanted in the brain
  Arms: Stimulation
Device: Direct Cortical Stimulation Sham — Sham trials where no electric pulse is delivered
  Arms: Sham

SUMMARY:
Purpose: To investigate whether rhythmic direct electrical stimulation (DES) causes entrainment of endogenous neural oscillatory activity and whether such activity improve cognition.

Participants: Drug-resistant epilepsy patients undergoing epilepsy surgery cortical mapping with continuous electrocorticography (ECoG) with intracranial electrodes.

Procedures (methods): Rhythmic electrical stimulation will be delivered via intracranial electrodes during routine extra-operative cortical mapping. Long-term ECoG, Pre-stimulation ECoG, peri-stimulation ECoG, and post-stimulation ECoG data will be analyzed to assess for entrainment of neural oscillations.

DETAILED DESCRIPTION:
The aim of this study is to characterize the entrainment of endogenous neural oscillatory activity using direct electrical stimulation (DES) of the brain and understand the effects on cognition.

In this study, the investigators will apply rhythmic DES to patients who are undergoing routine DES for cortical mapping as a part of their epilepsy surgery evaluation with the aim of entraining cortical neural oscillations at specific frequencies relevant to cognitive processing and neuropsychiatric disease. The investigators hypothesize that rhythmic DES within a naturally occurring oscillatory frequency will cause entrainment at that frequency (e.g. 10Hz rhythmic DES will entrain a 10 Hz alpha oscillation). Also, the investigators posit that rhythmic DES at the theta (5Hz), alpha(10Hz), and gamma (50Hz) frequencies will cause enhancement of neural oscillations in the gamma band.

The study follows a within-participant crossover design. Participants will perform one of the tasks described below and each task consists of multiple trials of varying difficulty. Stimulation will be applied concurrently through electrodes implanted for clinical determination of seizure focus. Equal number of stimulation and sham trials will be pseudo-randomly interleaved to get a balanced design (balanced across trial difficulty and trial type).

The investigators will apply electrical stimulation in the form of pulse trains. The applied electrical stimulation intensity, duration and frequency follow the parameters used for clinical assessments of language and seizure focus and fall below the clinically approved limits.

The investigators will measure participants performance on a simple working memory task during the above-described cortical electrical stimulation protocol. Alternately, participants can perform a face recognition task.

ELIGIBILITY:
Inclusion Criteria:

1. History of medically intractable epilepsy
2. Capable of giving informed consent
3. Aged 18 - 80 years, either sex

Exclusion Criteria:

1. Past or current history of other neurological illnesses including ischemic stroke, intracerebral hemorrhage, brain neoplasm.
2. Major systemic illness
3. Severe cognitive impairment defined as mini-mental state examination of less than 20
4. Severe psychiatric illness
5. Excessive use of alcohol or other substances

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Working Memory Task Performance - Accuracy | 1 Hour
  In this task, a sequence of items (alphabets or numerals) is presented followed by a delay. Following this, a single item which may or may not have been in the sequence is presented and the subject will be asked to indicate whether the item was in the previously presented sequence. A total of 150 trials will be performed with randomly interleaved sham trials where no stimulation is applied. Accuracy will be quantified in percentage correct.
Working Memory Task Performance - Reaction Time | 1 Hour
  In this task, a sequence of items (alphabets or numerals) is presented followed by a delay. Following this, a single item which may or may not have been in the sequence is presented and the subject will be asked to indicate whether the item was in the previously presented sequence. A total of 150 trials will be performed with randomly interleaved sham trials where no stimulation is applied. Reaction times will be quantified in milliseconds.

SECONDARY OUTCOMES:
Intracranial EEG | Intracranial EEG will be collected simultaneously when the participants perform the task. 1 Hour
  Spectral analysis and functional connectivity analysis of electrophysiology data will be performed using methods like multi-taper fft, wavelets, phase locking, Granger causality etc. The measures will be compared between sham and stimulation trials to identify if stimulation enhances neuronal entrainment. The correlation between the measures described above and the task performance will also be estimated.

OTHER OUTCOMES:
Facial Recognition Task Performance - Accuracy | 1 Hour
  Participants who consent will be administered this task. On a given trial, participants will be presented with images of two faces side-by-side. The faces will either match in terms of emotion category (e.g., 2 anger faces) or not (e.g., an anger face and a fear face). Faces presented together will always be of the same gender but different identities. Participants will be asked to determine whether the two faces presented depict the same emotion category. Participants will have 5 seconds to make the decision and indicate by pressing a key in the keyboard. Accuracy will be quantified in percent correct.
Facial Recognition Task Performance - Reaction Time | 1 Hour
  Participants who consent will be administered this task. On a given trial, participants will be presented with images of two faces side-by-side. The faces will either match in terms of emotion category (e.g., 2 anger faces) or not (e.g., an anger face and a fear face). Faces presented together will always be of the same gender but different identities. Participants will be asked to determine whether the two faces presented depict the same emotion category. Participants will have 5 seconds to make the decision and indicate by pressing a key in the keyboard. Reaction times will be quantified in milliseconds.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Frohlich, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Hae Won Shin, MD, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: Yes
De-identified electrophysiology data and task information (e.g. timing of each trial, timing of responses) will be shared at the end of the study in a central repository (e.g. zenodo)

REFERENCES:
- [Background] Alagapan S, Schmidt SL, Lefebvre J, Hadar E, Shin HW, Frӧhlich F. Modulation of Cortical Oscillations by Low-Frequency Direct Cortical Stimulation Is State-Dependent. PLoS Biol. 2016 Mar 29;14(3):e1002424. doi: 10.1371/journal.pbio.1002424. eCollection 2016 Mar. PMID 27023427
- Available data/document: Summary Data Set — http://dx.doi.org/10.5281/zenodo.45811 — Dataset supporting Alagapan et al. 2016 PLoS Biology